## Official title: HEMODYNAMIC CHANGES IN LEFT AND RIGHT LATERAL POSITION DURING ONE LUNG VENTILATION

Date: 01/05/2025

## NATIONAL AND KAPODISTRIAN UNIVERSITY OF ATHENS MEDICAL SCHOOL 2nd UNIVERSITY DEPARTMENT OF ANESTHESIOLOGY "ATTIKON" UNIVERSITY GENERAL HOSPITAL

| <b>Patient Consent Form</b> | |
|---|---|
| informed by the Anesthes<br>asked to participate, which<br>left and right lateral positive<br>study. The anesthetic tech | iologist about the nature of the study in which I am being h concerns the investigation of hemodynamic factors in the ions during one-lung ventilation, agree to participate in this iniques to be used are appropriate for this specific case, and be administered are approved by the National Organization |
| Helsinki for conducting me competent scientific bodie | I that the above study takes into account the Declaration of<br>nedical research on humans, that it has been approved by the<br>es of the hospital, and that it is completely safe for me.<br>on of personal data is ensured. |
| In light of all the above, I | agree to participate in the research. |
| | Date/ |
| The Patient | The Responsible Anesthesiologist |